CLINICAL TRIAL: NCT01128192
Title: Phase 2, Double-Blind, Randomized, Single Center Trial to Assess the Mechanism(s) Responsible for the Effect of the Somatostatin Analogue SOM230 (Pasireotide) in Healthy Male Volunteers. Version #2 05/09/2009
Brief Title: Somatostatin Analogue SOM230 (Pasireotide) in Healthy Male Volunteers
Acronym: Pasireotide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Robert R. Henry, MD (Other)
Collaborators: Veterans Medical Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Robert R. Henry, MD, Study Principal Investigator, Veterans Medical Research Foundation
Organization: Veterans Medical Research Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOM230Novartis/VMRF
Record Dates: First submitted 2009-09-15; First posted 2010-05-21 (Estimated); Results first posted 2014-12-25 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-12

CONDITIONS: Hyperglycemia
MeSH Terms: conditions — Hyperglycemia | interventions — pasireotide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pasireotide 600 µg sc bid (Experimental): n=19. Pasireotide 600 µg sc bid
  Interventions: Drug: pasireotide
- Pasireotide 900 µg sc bid (Experimental): n=19. Pasireotide 900 µg sc bid
  Interventions: Drug: pasireotide
- Pasireotide 1200 µg sc bid (Experimental): n=7. Due to increased severity of gastro-intestinal side effects, this arm was discontinued. These participants were only included in the safety analysis.
  Interventions: Drug: pasireotide

INTERVENTIONS:
Drug: pasireotide — Pasireotide 600 μg (batch number Y050DE) or 900 μg bid (batch number Y1270908) for subcutaneous injection. Placebo (batch number Y069HC) for subcutaneous injection.
  Other Names: SOM230

SUMMARY:
This clinical study will attempt to find out why in early studies in healthy volunteers, injections under the skin of pasireotide were associated with temporary increases in both fasting and post-meal glucose levels, along with possible increases in insulin and glucagon levels. Glucose refers to the amount of sugar in your blood and insulin and glucagon levels are amounts of hormones that lower and raise blood sugar.

The purpose of the study is to evaluate the effects of pasireotide on insulin resistance and secretion. Insulin is a natural hormone made by the pancreas (a gland inside the abdomen) that controls the level of sugar in the blood. Insulin permits cells to use sugar for energy. Insulin resistance is the condition in which higher than normal amounts of insulin are necessary to allow the sugar to enter the cells. Insulin secretion refers to the amount of insulin produced by the body and released in the blood. Glucagon is a hormone (chemical substance produced by the pancreas gland in the body) which increases blood glucose.

DETAILED DESCRIPTION:
This was a Phase 2, double-blinded, single-center study to assess the effects of pasireotide on insulin secretion and glucose metabolism in healthy male volunteers. Subjects who had given written informed consent and had been shown to satisfy the inclusion and exclusion criteria underwent baseline tests. An oral glucose tolerance test (OGTT) was administered on Day 1. If the OGTT results confirmed normal glycemia, the subject continued with baseline testing on Day 2 (2-step hyperglycemic clamp test with arginine stimulation) and Day 3 (2-step hyperinsulinemic euglycemic clamp (HEC) test with [3-3H]glucose). Each subject was then randomized into 1 of 3 dose groups: 600 µg twice daily (bid) delivered subcutaneously , pasireotide 900 µg bid delivered subcutaneously, or pasireotide 1200 µg bid delivered subcutaneously. Subcutaneous injections of pasireotide were given twice daily from Days 3-10 (for 8 consecutive days, starting from the evening of Day 3 and up to the morning injection on Day 10). On Study Days 8-10, the last 3 days of treatment with the pasireotide injections, the tests performed at Baseline (ie, the OGTT; the 2-step hyperglycemic clamp test with arginine stimulation; and the 2-step HEC test with [3-3H] glucose) were repeated. Subjects returned for a post-study safety follow-up visit 5 to 7 days after the last injection of the study drug and an H&P and safety labs (including a fasting glucose level) was performed. In addition, depending on subject convenience, a 3rd OGTT was either performed on this visit or was performed on another occasion convenient for subjects, in order to confirm that subjects' OGTT status had returned to baseline levels.

This additional post-study OGTT was added in a protocol amendment. Those subjects who completed the clinical trial and the follow-up visit before the amendment was approved were contacted and asked to return for another follow-up visit. The optional post-study OGTT was voluntary and subjects could choose not to participate. In order to reduce the severity of gastrointestinal adverse events (AEs), the protocol was amended (while keeping the blind intact) on 08 December 2009 to discontinue the pasireotide 1200 µg bid arm. The randomization scheme was subsequently adjusted to assign subjects in a 1:1 ratio to the 2 remaining arms: pasireotide 600 µg bid and pasireotide 900 µg bid.

ELIGIBILITY:
Inclusion Criteria:

* Lean, healthy, non-diabetic male.

Exclusion Criteria:

* Family history of diabetes, BMI over 25.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2009-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert R Henry, MD, Principal Investigator — Veterans Medical Research Foundation
Locations (1):
- CMR Center for Metabolic Research VASDHS, San Diego, California, United States

REFERENCES:
- [Result] Henry RR, Ciaraldi TP, Armstrong D, Burke P, Ligueros-Saylan M, Mudaliar S. Hyperglycemia associated with pasireotide: results from a mechanistic study in healthy volunteers. J Clin Endocrinol Metab. 2013 Aug;98(8):3446-53. doi: 10.1210/jc.2013-1771. Epub 2013 Jun 3. PMID 23733372
- See also: Study site Web site — http://www.vacmr.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy men aged 18-50 years with a body mass index (BMI) ≤25 kg/m2 who came to the VA San Diego Healthcare System Metabolic Research medical clinic. Recruitment occurred between August of 2009 until March 2010.
Pre-assignment Details: Participants were excluded if they had a family history of diabetes or a baseline diagnosis of impaired glucose tolerance.
Groups:
- Pasireotide 600 μg sc Bid: 19 healthy male volunteers were randomized to receive Pasireotide 600 μg (n=19). All participants completed the study.
- Pasireotide 900 μg sc Bid: 19 healthy male volunteers were randomized to receive Pasireotide 900 μg (n=19). All participants completed the study.
- Pasireotide 1200 μg sc Bid: 7 healthy male volunteers were randomized to receive Pasireotide 1200 μg (n=7). This arm was used in safety analysis only.
Period: Overall Study
Arm/Group | Pasireotide 600 μg sc Bid | Pasireotide 900 μg sc Bid | Pasireotide 1200 μg sc Bid
Started | 19 | 19 | 7
Completed | 19 | 19 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Nondiabetic males, aged 18-50 years with body mass index (BMI) ≤ 25. Subjects were not to have any family history of diabetes and no diagnosis of impaired glucose tolerance or gallstone disease.
Groups:
- Pasireotide 600 μg sc Bid: Pasireotide 600 μg sc bid n=19
- Pasireotide 900 μg sc Bid: Pasireotide 900 μg sc bid n=19
- Total: Total of all reporting groups
Arm/Group | Pasireotide 600 μg sc Bid | Pasireotide 900 μg sc Bid | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (4.6) | 24.6 (6.1) | 24.45 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Nondiabetic males, aged 18-50 years with body mass index (BMI) ≤ 25. Subjects were not to have any family history of diabetes and no diagnosis of impaired glucose tolerance or gallstone disease.
  Participants
    Female | 0 | 0 | 0
    Male | 19 | 19 | 38
Body Mass Index BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 23.30 (1.61) | 23.68 (2.04) | 23.49 (1.85)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 75.67 (8.11) | 74.49 (8.41) | 75.08 (8.26)

OUTCOME MEASURES:

1. Secondary Outcome: Change in Fasting Plasma Glucose Level
Description: An Oral Glucose Tolerance Test was performed at Day 1 (baseline) and Day 8 (post-treatment). Samples were taken at
  -30 min to assess the fasting plasma glucose level. The mean change in fasting plasma glucose level from Day 1 to Day 8 was assessed.
Time Frame: -30 minutes on Day 1 and -30 minutes on Day 8
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Pasireotide 600 µg sc Bid: Pasireotide 600 µg was injected subcutaneously twice daily from Day 3-10. Baseline OGTT was conducted on Day 1 (pre-treatment) and a post-treatment OGTT was conducted on Day 8.
- Pasireotide 900 µg sc Bid: Pasireotide 900 µg was injected subcutaneously twice daily from Day 3-10. Baseline OGTT was conducted on Day 1 (pre-treatment) and a post-treatment OGTT was conducted on Day 8.
Arm/Group | Pasireotide 600 µg sc Bid | Pasireotide 900 µg sc Bid
Number analyzed (Participants) | 19 | 18
mmol/L | -0.10 (0.36) | 0.12 (0.50)
Statistical Analysis 1: Comparison: Pasireotide 600 µg sc Bid; Change in fasting plasma glucose level; Test type: Superiority or Other; p = 0.240, ANOVA — Two sided P value
Statistical Analysis 2: Comparison: Pasireotide 900 µg sc Bid; Change in fasting plasma glucose level; Test type: Superiority or Other; p = 0.339, ANOVA — Two sided P value

2. Secondary Outcome: Change in Area Under the Curve (AUC) of Plasma Glucose 0-30mins, 30-180mins, 0-180mins During Oral Glucose Tolerance Test (OGTT)
Description: Blood samples were taken at -30 min, 0 min, 30 min, 60 min, 90 min, 120 min, 150 min, 180 min to assess the plasma glucose level. The mean change in plasma glucose level from Day 1 to Day 8 were calculated as Values on Day 8 - Values on Day 1.
Time Frame: 0-30 mins, 30-180 mins, 0-180 mins (Day 1 and Day 8)
Measure: Mean (Standard Deviation); unit: h*mmol/L
Arm/Group | Pasireotide 600 µg sc Bid | Pasireotide 900 µg sc Bid
Number analyzed (Participants) | 19 | 18
h*mmol/L
  AUC 0-30 min | -0.43 (0.43) | -0.86 (0.45)
  AUC 30-180 min | 14.72 (4.23) | 12.35 (4.25)
  AUC 0-180 min | 14.29 (4.02) | 11.49 (4.49)
Statistical Analysis 1: Comparison: Pasireotide 600 µg sc Bid; Pre and Post treatment Area Under the Curve (AUC) 0-30 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — Two sided P value
Statistical Analysis 2: Comparison: Pasireotide 600 µg sc Bid; Pre and Post treatment Area Under the Curve (AUC) 30-180 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — Two sided P Value
Statistical Analysis 3: Comparison: Pasireotide 600 µg sc Bid; Pre and Post treatment Area Under the Curve (AUC) 0-180 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — Two sided P Value
Statistical Analysis 4: Comparison: Pasireotide 900 µg sc Bid; Pre and Post treatment Area Under the Curve (AUC) 0-30 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — Two sided P value
Statistical Analysis 5: Comparison: Pasireotide 900 µg sc Bid; Pre and Post treatment Area Under the Curve (AUC) 30-180 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — Two sided P value
Statistical Analysis 6: Comparison: Pasireotide 900 µg sc Bid; Pre and Post treatment Area Under the Curve (AUC) 0-180 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — Two sided P value

3. Secondary Outcome: Change Fasting Plasma Insulin Level
Description: An Oral Glucose Tolerance Test was performed at Day 1 (baseline) and Day 8 (post-treatment). Samples were taken at -30 min to assess the fasting plasma insulin level. The mean change in fasting plasma insulin level from Day 1 to Day 8 was assessed.
Time Frame: -30 minutes on Day 1 and -30 minutes on Day 8
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Pasireotide 600 µg sc Bid | Pasireotide 900 µg sc Bid
Number analyzed (Participants) | 19 | 18
pmol/L | -6.62 (11.17) | -11.69 (10.96)
Statistical Analysis 1: Comparison: Pasireotide 600 µg sc Bid; Change in fasting plasma insulin level; Test type: Superiority or Other; p = 0.019, ANOVA — Two sided P value
Statistical Analysis 2: Comparison: Pasireotide 900 µg sc Bid; Change in fasting plasma insulin level; Test type: Superiority or Other; p < 0.001, ANOVA — Two sided P value

4. Secondary Outcome: Change in Area Under the Curve (AUC) of Plasma Insulin 0-30mins, 30-180mins, 0-180mins During Oral Glucose Tolerance Test (OGTT)
Description: Blood samples were taken at -30 min, 0 min, 30 min, 60 min, 90 min, 120 min, 150 min, 180 min to assess the plasma insulin level. The mean change in plasma insulin level from Day 1 to Day 8 were calculated as Values on Day 8 - Values on Day 1
Time Frame: 0-30 mins, 30-180 mins, 0-180 mins (Day 1 and Day 8)
Measure: Mean (Standard Deviation); unit: h*pmol/L
Arm/Group | Pasireotide 600 µg sc Bid | Pasireotide 900 µg sc Bid
Number analyzed (Participants) | 19 | 18
h*pmol/L
  AUC 0-30 min | -104.18 (90.60) | -100.90 (68.99)
  AUC 30-180 min | -184.96 (126.57) | -262.15 (158.58)
  AUC 0-180 min | -289.14 (162.54) | -363.06 (191.58)
Statistical Analysis 1: Comparison: Pasireotide 600 µg sc Bid; Pre and Post treatment Area Under the Curve (AUC) 0-30 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — Two sided P value
Statistical Analysis 2: Comparison: Pasireotide 600 µg sc Bid; Pre and Post treatment Area Under the Curve (AUC) 30-180 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — Two sided P value
Statistical Analysis 3: Comparison: Pasireotide 600 µg sc Bid; Pre and Post treatment Area Under the Curve (AUC) 0-180 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — Two sided P value
Statistical Analysis 4: Comparison: Pasireotide 900 µg sc Bid; Pre and Post treatment Area Under the Curve (AUC) 0-30 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — Two sided P value
Statistical Analysis 5: Comparison: Pasireotide 900 µg sc Bid; Pre and Post treatment Area Under the Curve (AUC) 30-180 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — Two sided P value
Statistical Analysis 6: Comparison: Pasireotide 900 µg sc Bid; Pre and Post treatment Area Under the Curve (AUC) 0-180 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — Two sided P value

5. Primary Outcome: Change in Insulin Basal Level
Description: Change from Day 2 and Day 9 of insulin basal levels (2-step hyperglycemic clamp test with arginine stimulation)
Time Frame: -30 min and -15 min on Day 2 and Day 9
Measure: Mean (Standard Deviation); unit: pmol/L
Groups:
- Pasireotide 600 µg sc Bid: Pasireotide 600 µg was injected subcutaneously twice daily from Day 3-10. Baseline hyperglycemic clamp test was conducted on Day 2 (pre-treatment) and a post-treatment hyperglycemic clamp was conducted on Day 9.
- Pasireotide 900 µg sc Bid: Pasireotide 900 µg was injected subcutaneously twice daily from Day 3-10. Baseline hyperglycemic clamp test was conducted on Day 2 (pre-treatment) and a post-treatment hyperglycemic clamp was conducted on Day 9.
Arm/Group | Pasireotide 600 µg sc Bid | Pasireotide 900 µg sc Bid
Number analyzed (Participants) | 19 | 19
pmol/L | -24.37 (10.42) | -29.60 (16.05)
Statistical Analysis 1: Comparison: Pasireotide 600 µg sc Bid; Change in Baseline Insulin Level; Test type: Superiority or Other; p < 0.001, ANOVA — Two sided P value
Statistical Analysis 2: Comparison: Pasireotide 900 µg sc Bid; Change in Baseline Insulin Level; Test type: Superiority or Other; p < 0.001, ANOVA — Two sided P value

6. Primary Outcome: Change in Area Under the Curve (AUC) of Plasma Insulin Level 0-10mins, 10-180mins, 0-180mins During Hyperglycemic Clamp
Description: Blood samples were taken at -30 min, -15 min, 0 min, 15 min, 30 min, 45 min, 60 min, 75 min, 90 min, 105 min, 120 min, 135 min, 150 min, 165 min, 180 min to assess the plasma insulin levels during Hyperglycemic Clamp (2-step hyperglycemic clamp test with arginine stimulation). The mean change in plasma insulin levels from Day 2 to Day 9 were calculated as Values on Day 9 - Values on Day 2.
Time Frame: 0-10 mins, 10-180 mins, 0-180 mins (Day 2 and Day 9)
Measure: Mean (Standard Deviation); unit: h*pmol/L
Arm/Group | Pasireotide 600 µg sc Bid | Pasireotide 900 µg sc Bid
Number analyzed (Participants) | 19 | 19
h*pmol/L
  AUC 0-10 min | -28.07 (19.15) | -27.95 (18.56)
  AUC 10-180 min | -1450.59 (1237.44) | -1474.65 (1009.00)
  AUC 0-180 min | -1478.65 (1254.66) | -1502.60 (1022.33)
Statistical Analysis 1: Comparison: Pasireotide 600 µg sc Bid; Pre and Post treatment Area Under the Curve (AUC) 0-10 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — Two sided P value
Statistical Analysis 2: Comparison: Pasireotide 600 µg sc Bid; Pre and Post treatment Area Under the Curve (AUC) 10-180 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — Two sided P value
Statistical Analysis 3: Comparison: Pasireotide 600 µg sc Bid; Pre and Post treatment Area Under the Curve (AUC) 0-180 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — Two sided P value
Statistical Analysis 4: Comparison: Pasireotide 900 µg sc Bid; Pre and Post treatment Area Under the Curve (AUC) 0-10 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — Two sided P value
Statistical Analysis 5: Comparison: Pasireotide 900 µg sc Bid; Pre and Post treatment Area Under the Curve (AUC) 10-180 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — Two sided P value
Statistical Analysis 6: Comparison: Pasireotide 900 µg sc Bid; Pre and Post treatment Area Under the Curve (AUC) 0-180 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — Two sided P value

7. Primary Outcome: Change in Basal Endogenous Glucose Production (EGP)
Description: Change from Day 3 and Day 10 of Basal EGP (Hyperinsulinemic-Euglycemic Clamp)
Time Frame: Day 3 and Day 10
Measure: Mean (Standard Deviation); unit: mg/kg/min
Groups:
- Pasireotide 600 µg sc Bid: Pasireotide 600 µg was injected subcutaneously twice daily from Day 3-10. Baseline Hyperinsulinemic-Euglycemic Clamp was conducted on Day 3 (pre-treatment) and post-treatment on Day 10.
- Pasireotide 900 µg sc Bid: Pasireotide 900 µg was injected subcutaneously twice daily from Day 3-10. Baseline Hyperinsulinemic-Euglycemic Clamp was conducted on Day 3 (pre-treatment) and post-treatment on Day 10.
Arm/Group | Pasireotide 600 µg sc Bid | Pasireotide 900 µg sc Bid
Number analyzed (Participants) | 19 | 19
mg/kg/min | -0.041 (0.342) | 0.112 (0.308)
Statistical Analysis 1: Comparison: Pasireotide 600 µg sc Bid; Change in Basal EGP; Test type: Superiority or Other; p = 0.608, ANOVA — Two sided P value
Statistical Analysis 2: Comparison: Pasireotide 900 µg sc Bid; Change in Basal EGP; Test type: Superiority or Other; p = 0.132, ANOVA — Two sided P value

8. Primary Outcome: Change in Low Dose % Endogenous Glucose Production (EGP) Inhibition
Description: Change from Day 3 and Day 10 of low dose % EGP Inhibition (Hyperinsulinemic-Euglycemic Clamp)
Time Frame: Day 3 and Day 10
Measure: Mean (Standard Deviation); unit: percentage of EGP Inhibition
Arm/Group | Pasireotide 600 µg sc Bid | Pasireotide 900 µg sc Bid
Number analyzed (Participants) | 19 | 19
percentage of EGP Inhibition | -7.54 (23.47) | -6.28 (16.31)
Statistical Analysis 1: Comparison: Pasireotide 600 µg sc Bid; Change in Low-Dose % EGP Inhibition; Test type: Superiority or Other; p = 0.178, ANOVA — Two sided P value
Statistical Analysis 2: Comparison: Pasireotide 900 µg sc Bid; Change in Low-Dose % EGP Inhibition; Test type: Superiority or Other; p = 0.111, ANOVA — Two sided P value

9. Primary Outcome: Change in High Dose % Endogenous Glucose Production (EGP) Inhibition
Description: Change from Day 3 and Day 10 of high dose % EGP Inhibition (Hyperinsulinemic-Euglycemic Clamp)
Time Frame: Day 3 and Day 10
Measure: Mean (Standard Deviation); unit: percentage of EGP inhibition
Arm/Group | Pasireotide 600 µg sc Bid | Pasireotide 900 µg sc Bid
Number analyzed (Participants) | 19 | 19
percentage of EGP inhibition | -2.06 (15.65) | 0.00 (0.00)
Statistical Analysis 1: Comparison: Pasireotide 600 µg sc Bid; Change in high-dose % EGP Inhibition; Test type: Superiority or Other; p = 0.573, ANOVA — Two sided P value

10. Primary Outcome: Change in Low-Dose Glucose Disposal Rate (GDR)
Description: Change from Day 3 and Day 10 in Low-Dose Glucose Disposal Rate (GDR) during Hyperinsulinemic-Euglycemic Clamp.
Time Frame: Day 3 and Day 10
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | Pasireotide 600 µg sc Bid | Pasireotide 900 µg sc Bid
Number analyzed (Participants) | 19 | 19
mg/kg/min | -0.029 (2.230) | 0.791 (2.144)
Statistical Analysis 1: Comparison: Pasireotide 600 µg sc Bid; Change in Low-Dose Glucose Disposal Rate (GDR); Test type: Superiority or Other; p = 0.956, ANOVA — Two sided P value
Statistical Analysis 2: Comparison: Pasireotide 900 µg sc Bid; Change in Low-Dose Glucose Disposal Rate (GDR); Test type: Superiority or Other; p = 0.125, ANOVA — Two sided P value

11. Primary Outcome: Change in High-Dose Glucose Disposal Rate (GDR)
Description: Change from Day 3 and Day 10 in High-Dose Glucose Disposal Rate (GDR) during Hyperinsulinemic-Euglycemic Clamp.
Time Frame: Day 3 and Day 10
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | Pasireotide 600 µg sc Bid | Pasireotide 900 µg sc Bid
Number analyzed (Participants) | 19 | 19
mg/kg/min | 0.004 (2.051) | -0.027 (2.099)
Statistical Analysis 1: Comparison: Pasireotide 600 µg sc Bid; Change in High-Dose Glucose Disposal Rate (GDR); Test type: Superiority or Other; p = 0.993, ANOVA — Two sided P value
Statistical Analysis 2: Comparison: Pasireotide 900 µg sc Bid; Change in High-Dose Glucose Disposal Rate (GDR); Test type: Superiority or Other; p = 0.956, ANOVA — Two sided P value

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected in real time as reported by each study subject. The study Investigators' reviewed and evaluated each individually reported Adverse Event within one week of reporting (if not immediately upon report).
Description: The investigator provided a listing of each subject's AEs. The individual AEs that occurred in each subject were then identified using the Investigator's term and AE frequency was summarized by dose group and adverse event.
Groups:
- Pasireotide 600 μg sc Bid; Pasireotide 900 μg sc Bid; Pasireotide 1200 μg sc Bid: Forty-five healthy male volunteers were randomized to receive pasireotide 600 μg (n=19), 900 μg (n=19) or 1200 μg (n=7) sc bid. All participants completed the study. Due to an increased severity of gastrointestinal AEs in the 1200 μg bid arm, randomization to this dose was discontinued after seven participants had completed the 7 days of treatment. These participants were included in the safety analyses only.
Arm/Group | Pasireotide 600 μg sc Bid | Pasireotide 900 μg sc Bid | Pasireotide 1200 μg sc Bid
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/7
Other Adverse Events (participants affected / at risk) | 18/19 | 18/19 | 7/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pasireotide 600 μg sc Bid (N=19) | Pasireotide 900 μg sc Bid (N=19) | Pasireotide 1200 μg sc Bid (N=7)
Nausea (Gastrointestinal disorders) | 10 (10) | 10 (10) | 5 (5) — 10 subjects (53.6%) in the 600 µg sc bid arm. 10 subjects (53.6%) in the 900 µg sc bid arm. 5 subjects (71.4%) in the 1200 µg sc bid arm.
Abdominal Cramping (Gastrointestinal disorders) | 6 (6) | 9 (9) | 4 (4) — 6 subjects (31.6%) in the 600 µg sc bid arm. 9 subjects (47.4%) in the 900 µg sc bid arm. 4 subjects (57.1%) in the 1200 µg sc bid arm.
Loose Stools (soft stools) (Gastrointestinal disorders) | 5 (5) | 13 (13) | 2 (2) — 5 subjects (26.3%) in the 600 µg sc bid arm. 13 subjects (68.4%) in the 900 µg sc bid arm. 2 subjects (28.6%) in the 1200 µg sc bid arm.
Burning Sensation (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0) — 4 subjects (21.1%) in the 600 µg sc bid arm. 2 subjects (10.5%) in the 900 µg sc bid arm.
Diarrhea (Gastrointestinal disorders) | 3 (3) | 4 (4) | 1 (1) — 3 subjects (15.8%) in the 600 µg sc bid arm. 4 subjects (21.1%) in the 900 µg sc bid arm. 1 subjects (14.3%) in the 1200 µg sc bid arm.
Fatigue (General disorders) | 3 (3) | 0 (0) | 1 (1) — 3 subjects (15.8%) in the 600 µg sc bid arm. 1 subject (14.3%) in the 1200 µg sc bid arm.
Vomiting/emesis (Gastrointestinal disorders) | 2 (2) | 3 (3) | 3 (3) — 2 subjects (10.5%) in the 600 µg sc bid arm. 3 subjects (15.8%) in the 900 µg sc bid arm. 3 subjects (42.8%) in the 1200 µg sc bid arm.
Gas (Flatulence) (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0) — 1 subject (5.3%) in the 600 µg sc bid arm. 4 subjects (21.1%) in the 900 µg sc bid arm.
Injection site redness (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) — 2 subjects (10.5%) in the 600 µg sc bid arm. 2 subjects (10.5%) in the 900 µg sc bid arm.
Injection site stinging (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) — 2 subjects (10.5%) in the 600 µg sc bid arm. 2 subjects (10.5%) in the 900 µg sc bid arm.
Upper respiratory infection (common cold) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) — 1 subject (5.3%) in the 600 µg sc bid arm. 3 subjects (15.8%) in the 900 µg sc bid arm.
Frequent Stools (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — 1 subject (5.3%) in the 600 µg sc bid arm.
Impacted wisdom tooth (General disorders) | 1 (1) | 0 (0) | 0 (0) — 1 subject (5.3%) in the 600 µg sc bid arm.
Light colored stool (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — 1 subject (5.3%) in the 600 µg sc bid arm.
Pressure in gut (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — 1 subject (5.3%) in the 600 µg sc bid arm.
Stomach ache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — 1 subject (5.3%) in the 600 µg sc bid arm.
Stomach cramps (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — 1 subject (5.3%) in the 900 µg sc bid arm.
Stomach fullness (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — 1 subject (5.3%) in the 600 µg sc bid arm.
Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — 1 subject (5.3%) in the 900 µg sc bid arm.
Injection site bruise (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — 1 subject (5.3%) in the 900 µg sc bid arm.
Sleepiness (General disorders) | 0 (0) | 1 (1) | 0 (0) — 1 subject (5.3%) in the 900 µg sc bid arm.
Dizziness (General disorders) | 0 (0) | 0 (0) | 1 (1) — 1 subject (14.3%) in the 1200 µg sc bid arm.
Histamine-like reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) — 1 subject (14.3%) in the 1200 µg sc bid arm.
Sweating (General disorders) | 0 (0) | 0 (0) | 1 (1) — 1 subject (14.3%) in the 1200 µg sc bid arm.
Vasovagal reaction while voiding (General disorders) | 0 (0) | 2 (2) | 0 (0) — 2 subjects (10.5%) in the 900 µg sc bid arm.
Infiltration, left ACFf (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Procedural complication: 1 subject (5.3%) in the 900 µg sc bid arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No